CLINICAL TRIAL: NCT07110740
Title: A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Evaluate Bioequivalence After Dry-powder Inhalation of UIC202005 or UI009 in Healty Volunteers
Brief Title: Bioequivalence Study Between UI009 and UIC202005 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI009-103
Record Dates: First submitted 2025-07-21; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UI009 (Experimental)
  Interventions: Drug: UI009
- UIC202005 (Active Comparator)
  Interventions: Drug: UIC202005

INTERVENTIONS:
Drug: UI009 — inhale UI009 twice a day on Day 1 and Day 8.
  Arms: UI009
Drug: UIC202005 — inhale UIC202005 twice a day on Day 1 and Day 8.
  Arms: UIC202005

SUMMARY:
A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Evaluate Bioequivalence After Dry-powder Inhalation of UIC202005 or UI009 in Healty Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 19 years or older at the time of screening.
2. Subjects whose body weight is at least 55 kg and with a body mass index (BMI) between 18.0 and 30.0 kg/m².
3. Subjects confirmed as healthy based on screening tests including vital signs, laboratory tests (hematology, biochemistry, urinalysis), and electrocardiogram (ECG), performed within 28 days prior to the first administration of the investigational product.
4. Female subjects who are not pregnant or breastfeeding, and who do not plan to become pregnant or breastfeed within 7 days after the last administration of the investigational product.
5. Subjects without congenital or chronic disease, and with no clinical significance based on physical examination.
6. Subjects who agree not to donate sperm (for males) or ova (for females), and whose partners agree to use medically acceptable contraception from the first administration to 7 days after the last dose.
7. Subjects able to read and understand a written informed consent, and willing to participate in the study.

Exclusion Criteria:

1. Subjects with any of the following medical histories or conditions deemed by the investigator to potentially interfere with the study:

   * Hypersensitivity to components of the investigational product or to other drugs such as aspirin or antibiotics
   * Hypersensitivity to sympathomimetic agents
   * hypersensitivity to inhaled lactose (allergic), galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
   * Cardiovascular disorders
   * Infectious respiratory diseases, especially tuberculosis or suspected infectious chronic obstructive pulmonary disease
   * Moderate to severe bronchiectasis
   * Asthma or COPD requiring emergency treatment
   * Hypokalemia
   * Hepatic dysfunction
   * Hyperthyroidism
   * Seizure disorders
2. Subjects with a history of taking or currently taking medications deemed by the investigator to potentially interfere with the study

   * Drugs known to interact with the investigational product or related drug classes (e.g., CYP3A4 inhibitors, beta-adrenergic agents, catecholamines, steroids, diuretics)
   * Enzyme-inducing or enzyme-inhibiting drugs (e.g., barbiturates) taken within 1 month prior to the first administration of the investigational product
   * Any prescription drugs taken within 10 days prior to the first administration of the investigational product
   * Any over-the-counter medications, including health supplements, herbal medicines, or dietary supplements, taken within 10 days prior to the first administration
3. Subjects who meet any of the following criteria during screening (including re-tests), and are deemed by the investigator to have clinically significant findings

   * Systolic blood pressure < 90 mmHg or > 140 mmHg
   * Diastolic blood pressure < 55 mmHg or > 90 mmHg
   * AST (GOT) or ALT (GPT) > 2.0 × upper limit of reference range
   * Serum potassium below the lower limit of the reference range
   * TSH below the lower limit of the reference range
   * FEV₁ or FEV₁/FVC outside the reference range
   * Positive results for serum tests: RPR Ab, HIV Ag/Ab, HBs Ag, HCV Ab
   * Positive result for any drug of abuse in the urine drug screening
4. Subjects who donated whole blood within 8 weeks, donated blood components within 4 weeks, or received a blood transfusion within 4 weeks prior to the first administration of the investigational product, or who plan to do so during the study period.
5. Subjects who consumed more than 5 cups/day (1 cup = 250 mL) of grapefruit-containing or caffeine-containing products within 3 months prior to the first administration, or who are unable to abstain from such consumption from 72 hours prior to dosing until the last pharmacokinetic blood sampling of each period.
6. Subjects who consumed more than 210 g/week of alcohol within 3 months prior to the first administration of the investigational product, or who are unable to abstain from alcohol from 72 hours prior to dosing until the last pharmacokinetic blood sampling of each period.
7. Subjects who smoked more than 10 cigarettes/day within 3 months prior to the first administration of the investigational product, or who are unable to abstain from smoking from 72 hours prior to dosing until the last pharmacokinetic blood sampling of each period.
8. Subjects who participated in another clinical trial and received an investigational drug within 6 months prior to the first administration (based on the last dosing date in the previous trial).
9. Subjects who are unable to consume the standard meals provided by the study center.
10. Subjects who are deemed by the investigator to be otherwise unsuitable for participation in the study for reasons not covered by the above exclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Cmax of Fluticasone propionate | Day 1 and Day 8: 0, 0.017, 0.033, 0.067, 0.1, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 hr
  Cmax(maxium concentration)
AUClast of Fluticasone propionate | Day1 and Day8: 0, 0.017, 0.033, 0.067, 0.1, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36hr
  Area under the curve to the last measurable concentration
AUC0.5hr of Salmeterol | Day1 and Day8: 0, 0.17, 0.033, 0.067, 0.1, 0.167, 0.333, 0.5hr
  Area under the curve from time 0 to 0.5 hours
AUClast of salmeterol | Day1 and Day8: 0, 0.017, 0.033, 0.067, 0.1, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36hr
  Area under the curve to the last measurable concentration
Cmax of Salmeterol | Day1 and Day8: 0, 0.017, 0.033, 0.067, 0.1, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36hr
  Cmax(maxium concentration)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided